CLINICAL TRIAL: NCT05983211
Title: A Biomarker-Directed Neuromodulation Trial Using Quantitative and Repetitive Transcranial Magnetic Stimulation in Amyotrophic Lateral Sclerosis (The QuARTS-ALS Trial)
Brief Title: Quantitative and Repetitive TMS in ALS - Recruiting for Stage 2
Acronym: QuARTS-ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QuARTS ALS
Record Dates: First submitted 2023-07-11; First posted 2023-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Repetitive transcranial magnetic stimulation; Corticospinal Excitability; Motor Neuron Disease; MR Spectroscopy; Cortical Hyperexcitability
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Stage 1 [Enrolment closed]:
  A prospective, single-arm, open-label pilot trial evaluating the safety, feasibility and changes in neuronal excitability biomarkers of accelerated rTMS using cTBS inhibitory paradigms over M1 in patients with ALS
  Stage 2 [CURRENTLY ENROLING]:
  A prospective, single-arm, open-label pilot trial evaluating the safety, target engagement via biomarkers, and dose discovery of multi-targeted, accelerated continuous theta burst stimulation (cTBS) regimen of repetitive transcranial magnetic stimulation (rTMS) over multiple primary motor cortex (M1) regions bilaterally with repeated maintenance cTBS sessions for 24 weeks in patients with ALS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated cTBS Neuromodulation (Experimental): Stage 2 [CURRENTLY ENROLLING]:
  ALS patients receiving an accelerated schedule of continuous theta burst rTMS bilaterally at multiple M1 regions at a regimen of 40 seconds, 1 minute 20 seconds, 2 minutes, or 4 minutes per treatment for up to 8 treatment sessions per day, delivered one per hour, over 5 days. Additional single-day maintenance treatments will follow these 5 days at a frequency of every 2 weeks for 12 weeks, then every 4 weeks for 12 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Stage 2 [CURRENTLY ENROLLING]:
  Accelerated rTMS using continuous theta burst stimulation (cTBS) inhibitory paradigms over bilateral M1 including hand, leg, and bulbar regions outputted at 90% of resting motor threshold, using bursts of 3 pulses at 50 Hz. Bursts are repeated at 5 Hz for a total of 600, 1200, 1800, or 3600 pulses over 40 seconds, 1 minute 20 seconds, 2 minutes, or 4 minutes. ALS patients will receive rTMS bilaterally for up to 8 treatment sessions per day, delivered one per hour, over 5 days, followed by single-day maintenance treatments at a frequency of every 2 weeks for 12 weeks, then every 4 weeks for 12 weeks.

SUMMARY:
Stage 1 [Enrolment closed]:

The goal of this open-label pilot clinical trial is to evaluate the safety and feasibility of accelerated, repetitive transcranial magnetic stimulation (rTMS) using continuous theta-burst stimulation (cTBS) in patients with ALS.

Stage 2 [CURRENTLY ENROLLING]:

The goal of this open-label pilot clinical trial is to evaluate the safety, tolerability and target engagement of accelerated, high dose cTBS using TMS in patients with ALS.

DETAILED DESCRIPTION:
Stage 1 [Enrolment closed]:

The purpose of this stage is to evaluate the safety, feasibility, and changes in neuronal excitability biomarkers of accelerated repetitive transcranial magnetic stimulation (rTMS) using continuous theta-burst stimulation (cTBS) inhibitory paradigms over M1 in patients with ALS.

Stage 2 [CURRENTLY ENROLLING]:

The purpose of this study is to:

1. Assess the safety and feasibility of accelerated cTBS treatment with maintenance cTBS treatments in individuals with ALS over a 24-week period.
2. Assess changes in MR spectroscopy measures of glutamate and GABA, ATP and metabolites markers, and neuronal structure markers, changes in serum neurofilament light chain, and changes in corticohyperexcitability biomarkers measured by single and paired pulse quantitative TMS.
3. Assess the changes in ALSFRS-R and muscle strength dynamometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with ALS as per the 2020 Gold Coast Criteria;
* Age ≥ 18 years;
* Able to provide informed consent to study procedures and treatments;
* Patients are allowed to start or continue the standard of care treatments for ALS. Presently these include oral riluzole, and oral or intravenous edaravone;
* Able to lie supine without BiPAP or breathing discomfort for at least 1 hour;
* No contraindications to TMS as follow;
* Metal implants in the head or neck (such as aneurysm clips, vessel stents), implanted medication pump, implanted brain stimulators, pacemaker, cochlear implants, or history of epilepsy. Dental fillings are permitted;
* Current use of medications or medical conditions that, at the discretion of the Principal Investigator, could potentially increase the risk of seizures or interfere with stage outcomes;
* On medications that affect TMS measures in a PRN regimen (as needed). Continuous use of these medications on a fixed dose of 30 days prior to first Baseline Visit or after a wash-out period of 2 weeks is accepted. These medications include, but are not limited to: benzodiazepines, muscle relaxants, tricyclic antidepressants, selective and non-selective serotonin reuptake inhibitors, hypnotics (including anti-histamine drugs) and anticholinergics drugs;
* History of seizure, convulsion, or epilepsy;

Exclusion Criteria:

* Known diagnosis of dementia;
* Definitely or possibly pregnant (if applicable);
* History of allergy to Ag-AgCl electrode gel (standard neurophysiology electrodes);
* Unable to tolerate TMS procedures;
* Lack of MRI brain performed prior to the stage, inability to perform an MRI at baseline due to orthopnea, or:
* Large body habitus and not fitting comfortably into the scanner;
* Difficulty laying still for up to 1 hour in the MRI unit or significant claustrophobia;
* Metallic implants;
* Any contraindications for receiving rTMS treatment as follow:
* have received rTMS for any previous indication due to the potential compromise of subject blinding;
* have increased intracranial pressure, a space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, significant head trauma with clear radiological evidence of cerebrovascular injury on imaging;
* have an intracranial implant or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
* have clinically significant laboratory abnormality, in the opinion of the one of the principal investigators or study physicians;
* are currently taking more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy;
* Any other clinical condition that, in the opinion of the Site Investigator, would place the subject at increased risk or preclude the subject's full compliance with completion of the stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of cTBS rTMS in patients with ALS | Up to 30 days before compared to during the initial 5 days of cTBS treatment and up to 24 weeks after
  Incidence of AEs and SAEs after accelerated continuous theta burst stimulation inhibitory intervention in individuals with ALS through the incidence of repetitive TMS treatment related adverse events, serious adverse events, and discontinuations due to adverse events/serious adverse events.

SECONDARY OUTCOMES:
Neurofilament light chain (NfL) levels | Up to 30 days before compared to the last treatment day, 12 weeks, and 24 weeks after cTBS treatment
  Change in concentration of serum neurofilaments from Baseline to Treatment, Week 12, and Week 24
ALSFRS-R scores | Up to 30 days before compared to 12 and 24 weeks after cTBS treatment
  >/= 6-point decline in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) scores from Baseline to Week 12 and Week 24. The ALSFRS-R measures functional ability in ALS with a minimum 0, maximum 48, and where a higher score means a better outcome.
Corticospinal Excitability change measured by quantitative TMS | Up to 30 days before compared to 12 and 24 weeks after cTBS treatment
  Change from baseline in Resting Motor Threshold (RMT), Cortical Silent Period (CSP), Short Intracortical Inhibition (SICI), and Short Intracortical Facilitation (SICF). All measurements use the same units.
Magnetic Resonance Spectroscopy parameters as measured by MRS | Up to 30 days before compared to the end of treatment week, 5 weeks, 12 weeks, and 24 weeks after cTBS treatment
  Change from baseline in Glutamate, GABA, neuronal and redox metabolite ratios. All measurements use the same units.

CONTACTS AND LOCATIONS:
Overall Officials: Agessandro Abrahao, Dr., Principal Investigator — Sunnybrook Health Sciences Centre; University of Toronto; Lorne Zinman, Dr., Principal Investigator — Sunnybrook Health Sciences Centre; University of Toronto; Sean Nestor, Dr., Principal Investigator — Sunnybrook Research Institute; University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No